CLINICAL TRIAL: NCT06293183
Title: The Effect of Artificial Intelligence Supported Mobile Learning Developed for Hemodialysis Patients on Nutrition/Fluid Intake Control and Individual Management
Brief Title: The Effect of Artificial Intelligence Supported Mobile Learning on Nutrition/Hydration Control and Individual Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sevda Tüzün Özdemir, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGE-HEM-STO-01
Record Dates: First submitted 2024-02-15; First posted 2024-03-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cronich Kidney Disease
Keywords: Hemodialysis; mobile learning; hydration; nutrition; nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): After the purpose and method of the research are explained, a written informed consent form will be obtained and the Patient Introduction Form will be filled out. Mobile phone usage skills of patients undergoing hemodialysis treatment will be evaluated using the Digital Literacy Scale. Individuals in the initiative group will be given individual training on how to use the application through the application demo. Individuals in the initiative group will be given consultancy by the researcher while downloading the application and logging in with their username. Questionnaires and scale forms will be applied to the patients in the control group on the 0th day, the 14th day, and at the 1st, 2nd and 3rd months. Laboratory values and intradialytic weight information will be obtained from patient files.
  Interventions: Other: Mobile app
- Control group (No Intervention): After the purpose and method of the research are explained, a written informed consent form will be obtained and the Patient Introduction Form will be filled out. No intervention will be made to the participants in this group. Questionnaires and scale forms will be applied to the patients in the control group on the 0th day, 14th day, 1st, 2nd and 3rd months. Laboratory values and intradialytic weight information will be obtained from patient files.

INTERVENTIONS:
Other: Mobile app — Participants in the intervention group will be expected to watch the training video in the mobile application installed on their phones or tablets and then regularly enter all the food and liquid amounts they consume during the day into this application. In the mobile application data entry area, visuals that will be included in the application showing the amount and types of foods consumed by the participants during the day (1 soup bowl, 1 vegetable dish plate, 1 meat dish plate, 1 water glass, 1 tea glass, tablespoon, dessert spoon, teaspoon, ladle). etc.) will choose through. The mobile application will calculate the total amount of liquid consumed by the participants in 24 hours, and will give a yellow warning when the amount of liquid consumed is 2-2.5 liters, an orange warning when it is 2.5-3 liters, and a red warning when it is 3 liters and above. This will contribute to reducing the amount of fluid intake of participants between two dialysis sessions.
  Arms: Intervention group

SUMMARY:
The adherence to recommended nutrition and fluid restrictions is crucial for the success of hemodialysis treatment. However, approximately 80% of patients receiving HD treatment are non-compliant with fluid restriction, leading to various complications. Cardiovascular complications are among the most common complications associated with this issue. When reviewing national and international literature on the subject, it is observed that in order to improve treatment adherence in HD patients, written materials are often used in addition to individual or group education sessions, focusing mainly on assessing patients' quality of life and self-efficacy. However, a mobile-supported learning method that enables patients to manage their nutrition and fluid control individually is not commonly utilized.

This research aims to investigate the impact of an artificial intelligence-supported mobile application developed for HD patients on the control of nutrition/fluid intake and individual management.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) in the late stage is defined as the progressive and irreversible loss of renal functions due to various reasons leading to a decrease in glomerular filtration rate (GFR). It is estimated that there are 37 million diagnosed cases of CKD worldwide, with CKD ranking ninth among the leading causes of death in the United States. Among the treatment options for end-stage renal failure are hemodialysis (HD), peritoneal dialysis (PD), and transplantation (TX), with HD being the most preferred method by patients. According to the 2022 registration data from the Turkish Society of Nephrology, there were a total of 86,665 CKD patients by the end of 2022, with 71.22% of these patients (n: 61,723) receiving HD treatment.

In patients undergoing HD treatment, the weight gained between two dialysis sessions is defined as interdialytic weight gain (IDWG). The development of hypervolemia due to excessive weight gain can lead to both systemic illnesses and problems during the treatment process. Particularly, cardiovascular problems rank first among systemic illnesses (43%), leading to complications related to excessive ultrafiltration (UF) during the treatment process (hypotension, muscle cramps, nausea-vomiting). Elevated IDWG generally leads to hypertension, left ventricular hypertrophy, pulmonary edema, congestive heart failure, and higher mortality rates due to all these cardiac problems. The ideal IDWG is expected to be in the range of 1-2 kg or 3-5%. In a study, it was reported that 85% of HD patients had an IDWG of >1.5 kg, especially young, male, and diabetic patients tend to have high IDWG, which leads to an increase in mortality rates due to cardiovascular diseases. Similar results have been reported in many other studies. According to estimates from the United States Renal Data System, cardiovascular events account for 40% of deaths. The 2022 data from the Turkish Society of Nephrology reports that cardiovascular diseases were the leading cause of death (46.3%) among HD patients in our country by the end of 2022. Similar results have been reported in many other studies.

The concept of individual management is defined as the ability of patients with a chronic disease to manage their illness, change their lifestyle, and therefore, live with a chronic disease. Individual management in HD patients requires various skills, including adherence to recommended treatment (e.g., weight gain, nutrition), effective symptom management, problem-solving ability, disease control, decision-making, and communication with the healthcare team. Therefore, increasing individual management in HD patients is known to be associated with increased treatment adherence and better clinical outcomes. In a study, it was found that a mobile application-based individual management program developed to determine the effects of HD patient role behaviors, basic psychological needs, and individual management was effective in increasing patients individual management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Conscious and able to communicate,
* Having received hemodialysis treatment for the last 3 months,
* Able to use an Android-based phone (for those who do not have a personal mobile phone, an application will be installed on the primary caregiver's phone),
* Having a digital literacy scale score over 17,
* Patients who agree to participate in the research will be included in the research.

Exclusion Criteria:

* Patients diagnosed with acute renal failure
* Having vision problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Fluid intake compliance | 4 months
  Nutrition (for nutrition, Nutritional Behavior Scale in Hemodialysis Patients score) and fluid intake compliance (for fluid compliance, Nutritional Behavior Scale in Hemodialysis Patients score) of the patients included in the study will be evaluated. In addition, the entry kilogram information of the patients participating in the study will be taken from the patient files before the dialysis session. .
  Fluid Control Scale in Hemodialysis Patients: It consists of a total of 24 items and three sub-dimensions (knowledge, behavior and attitude), the lowest score from the scale is 24 and the highest score is 72. As the score increases, patients' compliance with fluid control also increases.
  Nutritional Behavior Scale of Hemodialysis Patients: It was developed to evaluate the nutritional behavior of patients receiving hemodialysis treatment. The scale score is between 13-65. The higher the score, the more "good behavior" is considered.

SECONDARY OUTCOMES:
Change of individual management | 4 months
  Individual management of patients will be evaluated with the "Hemodialysis Self-Management Instrument (HDSMI-18)" scale.
  Individual Management Scale for Hemodialysis Patients: The tool measuring the individual management behaviors of hemodialysis patients was developed to evaluate the individual management behaviors of patients. The scale includes four subheadings and 20 items describing the patient's disease management behaviors in the last 3 months. Scale; It is a four-point Likert type ranging from never (1 point), rarely (2 points), sometimes (3 points) and always (4 points), and each item is rated with a total of 4 points. The total score range varies between 20-80, with higher scores indicating higher levels of individual management behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Daviva Buca Dialysis Centre, Izmir, Buca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When the study is completed and published, other researchers who will need research data will be able to contact me in case of any request.